CLINICAL TRIAL: NCT06526715
Title: Balance Effects of Morton´s Extension in Flat Foot. A Pre-post-test Study.
Brief Title: Balance Effects of Morton´s Extension in Flat Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Collaborators: Universidad de León (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist, profesor, Universidad Complutense de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/458-E
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subjects
Keywords: balance; Foot; Orthopedics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morton.s extension treatment (Experimental): Appliation of Morton´s extension treatment simulation
  Interventions: Other: Morton extension

INTERVENTIONS:
Other: Morton extension — A Morton extension with a height of 5 mm was insert from the proximal area of the first metatarsal head to the base of the proximal phalanx of the Hallux of the subjects' bare feet using a paper bandage. The material, shape, size, and thickness of the Morton Extension were the same.

SUMMARY:
The aim of this study is to simulate the orthopedic treatment called Morton's extension on flat foot patients to check balance effects in standing position.

DETAILED DESCRIPTION:
The objective of this study is to perform an assimilation of the orthopedic treatment called morton extension on flat foot patients to verify the balance with stabilometry study.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18 to 30 with flexible flat feet.

Exclusion Criteria:

* Participants who have had any previous limb surgery, and/or previous lower limb trauma within the last year
* Uncorrected hearing or visual impairment.
* Lumbar pathology with radicular involvement.
* Pregnancy.
* Healthy participants performing strenuous exercise.
* Diagnosed active or inactive rheumatic or inflammatory disease.
* Participants consuming alcohol within 24 hours prior to recording or stimulants 6 hours prior to testing (e.g. caffeine).
* Participants who have a history of injury with residual lower extremity symptoms within the past year.
* Participants with evidence of a leg length discrepancy (difference in distance from the anterior superior iliac spine to the superior iliac spine at the surface of the most prominent aspect of the medial malleolus) of more than 1 cm 19
* Having at least 15 degrees of ankle dorsiflexion.
* Participants with evidence of balance deficit, as determined through oral questioning about falls and by use of the Balance Evaluation Systems Test (BESTest).
* Participants with neurological pathology with lower limb deformities, sensory-motor disturbances, neuromuscular pathology, or neurovascular disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Length in millimetres of the centre of pressures. Untreated | Through study completion, an average of 4 days
  Length of the centre of pressures described in millimetres.
Area of the ellipse. Untreated | Through study completion, an average of 4 days
  Area of the ellipse in square millimeters.
Inclination of the ellipse in degrees.Untreated | Through study completion, an average of 4 days
  Inclination of the ellipse generated by the centre of pressures in 30 seconds in degrees.
Length-area ratio. Untreated | Through study completion, an average of 4 days
  Fraction of the length of the ellipse between the surface of the ellipse in millimetres.
Delta x. Untreated | Through study completion, an average of 4 days
  Displacement on the x-axis within the ellipse calculated from the movements of the barycentre. In millimetres.
Delta y. Untreated | Through study completion, an average of 4 days
  Displacement on the y-axis within the ellipse calculated based on the movements of the barycentre. In millimetres.
Displacement on the major axis or y-axis. Untreated | Through study completion, an average of 4 days
  Displacement in millimetres of the y-axis.
Displacement on the minor axis or x-axis. Untreated | Through study completion, an average of 4 days
  Displacement in millimetres of the y-axis.
Maximum oscillation. Untreated | Through study completion, an average of 4 days
  Measurement of the length in millimetres of the maximum oscillations.
Minimum oscillation in millimetres. Untreated | Through study completion, an average of 4 days
  Measurement of the length in millimetres of the minimum oscillations
Length in millimetres of the centre of pressures with treatment | Through study completion, an average of 4 days
  Length of the centre of pressures described in millimetres.
Area of the ellipse with treatment | Through study completion, an average of 4 days
  Area of the ellipse in square millimeters.
Inclination of the ellipse in degrees with treatment | Through study completion, an average of 4 days
  Inclination of the ellipse generated by the centre of pressures in 30 seconds in degrees.
Length-area ratio with treatment | Through study completion, an average of 4 days
  Fraction of the length of the ellipse between the surface of the ellipse in millimetres.
Delta x with treatment | Through study completion, an average of 4 days
  Displacement on the x-axis within the ellipse calculated from the movements of the barycentre. In millimetres.
Delta y with treatment | Through study completion, an average of 4 days
  Displacement on the y-axis within the ellipse calculated based on the movements of the barycentre. In millimetres.
Displacement on the major axis or y-axis with treatment | Through study completion, an average of 4 days
  Displacement in millimetres of the y-axis.
Displacement on the minor axis or x-axis with treatment | Through study completion, an average of 4 days
  Displacement in millimetres of the y-axis.
Maximum oscillation with treatment | Through study completion, an average of 4 days
  Measurement of the length in millimetres of the maximum oscillations.
Minimum oscillation in millimetres with treatment | Through study completion, an average of 4 days
  Measurement of the length in millimetres of the minimum oscillations

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Martínez Jiménez, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Eva María Martínez-Jiménez, León, Spain

IPD SHARING:
Plan to Share IPD: No